CLINICAL TRIAL: NCT00646828
Title: Cardiovascular Evaluation of a Rare Condition With Hyperaldosteronism Without Hypertension: PHA 1
Brief Title: Cardiovascular Evaluation of Adult PHA 1 Patients
Acronym: PHACARV
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P070139
Record Dates: First submitted 2008-02-28; First posted 2008-03-31 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2010-07

CONDITIONS: Pseudohypoaldosteronism Type 1
Keywords: Pseudohypoaldosteronism type 1; Mineralocorticoid receptor; Aldosterone; Cardiovascular disease
MeSH Terms: conditions — Pseudohypoaldosteronism; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- without PHA1: patients without mineralocorticoid receptor mutation
- PHA 1: patients with a rare disease, pseudohypoaldosteronism type 1, due to heterozygous inactivating mutations of the mineralocorticoid receptor

SUMMARY:
Vascular and cardiac alterations are associated with aldosterone effects are evidenced in experimental models and aldosterone receptor blockade is of clear benefit in cardiac disease (heart failure). The study aims at assessing vascular and cardiac alterations in adults with a chronic increase in circulating aldosterone without hypertension. The investigated population will be patients with a rare disease, pseudohypoaldosteronism type 1, due to heterozygous inactivating mutations of the mineralocorticoid receptor.

DETAILED DESCRIPTION:
The study includes adult patients with mineralocorticoid receptor mutation as compared with not affected relatives. It includes also relatives of adult relative of patients with PHA1 in whom no mutation was found. Cardiovascular evaluation is conducted with cardiac and vascular ultrasound assessment and cardiac NMR, ambulatory blood pressure measurement.

Protocol duration is 2 days . Detailed genetic study is conducted in family without identified mutation in MINERALORECEPTOR.

ELIGIBILITY:
Inclusion criteria:

* Age over 18
* Male or female gender
* Genotype in the PHA1.NET network

Exclusion criteria:

* Not membership to a regime of Social Security or to a CMU
* Against indication in the realization of a MRI
* Cardiac NMR not possible
* Known cardiovascular disease for person not carrying MR mutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient with Pseudohypoaldosteronism type 1 and the family of these patient who dont have mineralocorticoid receptor mutation
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Cardiac or vascular abnormality at ultrasound or NMR evaluation | day one

SECONDARY OUTCOMES:
Extracellular volume, biology, autonomic nervous system abnormality | day one + day two
New gene responsible for PHA1 | day one

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte ESCOUBET, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bichat, Paris, France

REFERENCES:
- [Background] Pujo L, Fagart J, Gary F, Papadimitriou DT, Claes A, Jeunemaitre X, Zennaro MC. Mineralocorticoid receptor mutations are the principal cause of renal type 1 pseudohypoaldosteronism. Hum Mutat. 2007 Jan;28(1):33-40. doi: 10.1002/humu.20371. PMID 16972228
- [Background] Sacre K, Brihaye B, Hyafil F, Serfaty JM, Escoubet B, Zennaro MC, Lidove O, Laissy JP, Papo T. Asymptomatic myocardial ischemic disease in antiphospholipid syndrome: a controlled cardiac magnetic resonance imaging study. Arthritis Rheum. 2010 Jul;62(7):2093-100. doi: 10.1002/art.27488. PMID 20506512
- [Derived] Escoubet B, Couffignal C, Laisy JP, Mangin L, Chillon S, Laouenan C, Serfaty JM, Jeunemaitre X, Mentre F, Zennaro MC. Cardiovascular effects of aldosterone: insight from adult carriers of mineralocorticoid receptor mutations. Circ Cardiovasc Genet. 2013 Aug;6(4):381-90. doi: 10.1161/CIRCGENETICS.113.000115. Epub 2013 Jul 14. PMID 23852419